CLINICAL TRIAL: NCT02851381
Title: Compassionate Single Subject Use of FG-3019 in Locally Advanced, Unresectable Pancreatic Cancer (Emergency Use of a Test Article)
Brief Title: Compassionate Single Subject Use of FG-3019 (FibroGen) in Locally Advanced, Unresectable Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient passed before treatment could be started
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-001170
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pamrevlumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FG-3019 (Other): Treatment of Pancreatic Cancer with FG-3019
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — The FG-3019 treatment will be administered over a 28-day cycle:
  * Dose: 35 mg/kg
  * Route: IV over one hour following completion of gemcitabine infusion
  * Schedule:
    * Days 1, 8, and 15
    * Please note that Day 8 infusion will on be completed during the first treatment cycle

SUMMARY:
Single compassionate use subject is an 83 year old woman with a history of lymph node positive breast cancer and recently diagnosed pancreatic cancer in May. With an Eastern Cooperative Oncology Group (ECOG) of 2, it is felt that she cannot tolerate more aggressive chemotherapy. The investigators propose to administer FG-3019 on a compassionate pleas basis in combination with gemzar. The patient is currently being treated and is tolerating gemzar.

DETAILED DESCRIPTION:
The FG-3019 treatment will be administered over a 28-day cycle:

* Dose: 35 mg/kg
* Route: IV over one hour following completion of gemcitabine infusion
* Schedule:

  * Days 1, 8, and 15
  * Please note that Day 8 infusion will on be completed during the first treatment cycle

On Drug Evaluation

The patient will be seen prior to every FG-3019 treatment by the treating physician. The following procedures will be conducted at each visit:

* History and thorough symptom assessment
* Physical examination
* Laboratory assessments (these can be collected up to 3 days prior to treatment):
* Complete blood count (CBC) and differential
* Comprehensive Metabolic Panel (Chemistry): bicarbonate, blood, urea, nitrogen (BUN), calcium, creatinine, glucose, potassium, sodium
* Liver Function Tests: Alkaline phosphatase (ALP), Alanine transaminase (ALT), Aspartate transaminase (AST), total bilirubin
* Carbohydrate antigen (CA) 19-9

ECGs will be conducted during the screening and end of treatment visits. CT scans of the chest and abdomen will be done every 12 to 16 weeks.

All of these data will be recorded and stored with their source documents.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent form
* Have adequate liver function
* Have adequate bone marrow function

Exclusion Criteria:

* History of allergy or hypersensitivity to human, humanized or chimeric monoclonal antibodies
* Any medical or surgical condition that may place the subject at increased risk while on treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with treatment requirements
* Current abuse of alcohol or drugs

Ages: 83 Years to 83 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
FG-3019 treatment regimen to increase OS (overall survival) | 7.7 months

CONTACTS AND LOCATIONS:
Overall Officials: John Glaspy, M.D., Principal Investigator — Professor of Medicine

IPD SHARING:
Plan to Share IPD: No